CLINICAL TRIAL: NCT05193799
Title: Monocentric, Open Study for the Evaluation of the Tolerance of Three Class I Medical Devices Under Dermatological Control.
Brief Title: Evaluation of the Tolerance of Three Masks Under Dermatological Control.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Kolmi Hopen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21E2022
Record Dates: First submitted 2021-12-22; First posted 2022-01-18 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Healthy Population

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Investigational device#1 = Kolmi® Op-AirTM KALM (Experimental)
  Interventions: Device: Investigational devices must be used 8 hours per day
- Investigational device#2 = Kolmi® Op-Air OneTM (Experimental)
  Interventions: Device: Investigational devices must be used 8 hours per day
- Investigatonal device#3 = Kolmi® Op Air-Pro® Oxygen (Experimental)
  Interventions: Device: Investigational devices must be used 8 hours per day

INTERVENTIONS:
Device: Investigational devices must be used 8 hours per day — During 3 consecutive days

SUMMARY:
This is a monocentric, open and randomized study. The purpose is to evaluate the cutaneous tolerance of three medical masks (class I medical device) after 3 consecutive days of use on a population with normal or sensitive skin.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Subject;
2. Sex: male or female ;
3. Age: more than 18 years ;
4. Phototype: I to IV on the Fitzpatrick scale;
5. For half of the population in each group : subject presenting a sensitive skin on the face confirmed by an interrogatory with the investigator (see Appendix 19.1).
6. Subjects who did not use any new cosmetic product on the face in the past 30 days and who agree not to change them during the study period.
7. Subject having given freely and expressly his/her informed consent;
8. For subjects randomized to group 3: Fit test FFP on M52014-WH

Exclusion Criteria:

In terms of population

1. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship;
2. Subject in a social or sanitary establishment;
3. Subject suspected to be non-compliant according to the investigator's judgment;
4. Subject enrolled in another clinical trial or which exclusion period is not over.
5. Subject majors under curatorship, safeguard of justice, activated future protection mandate or family authorization In terms of associated pathology
6. Subject with a condition or receiving a medication which, in the investigator's judgment, put the subject at undue risk;
7. Subject suffering from a severe or progressive disease.
8. Subject's with too many hairs, bears,(to put above) skin lesions, skin disease or severe acne on the face that could interfere with the tolerance evaluation.
9. Subject' who is allergic to one or several component of the studied devices. Relating to previous or ongoing treatment
10. Subject undergoing a topical treatment on the test area or a systemic treatment:

    * anti-inflammatory medication and/or antihistamines during the 2 weeks prior to screening and during the study;
    * corticosteroids during the 2 weeks and prior to screening and during the study;
    * retinoids and/or immunosuppressors during the 3 months prior to screening and during the study;
11. Subject having started or changed any hormonal treatment during the three previous months.

    In terms of lifestyle
12. Intensive exposure to sunlight or UV-rays within the previous month and/or foreseen during the study;
13. Subject planning to change her/his life habits during the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Cutaneous tolerance | Days 3
  Evaluation of the percentage of subjects presenting no relevant clinical or functional signs of cutaneous intolerance after 3 days of use of the three medical devices

SECONDARY OUTCOMES:
Subjective appreciation | 3 days
  Analysis of the subject's answer to a subjective evaluation questionnaire
Number of Adverse event | 3 days
  Collection of cutaneous and systemic Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: Siham Rharbaoui, Principal Investigator — Eurofins Dermscan Pharmascan
Locations (1):
- Laboratoire Eurofins Dermscan Pharmascan, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: Undecided